CLINICAL TRIAL: NCT05264389
Title: Post-market Clinical Follow-up (PMCF) Study of the Poly-Tape Devices for Medial Patellofemoral Ligament (MPFL) Reconstruction
Status: Recruiting | Type: Observational
Sponsor: Xiros Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CRE 022
Record Dates: First submitted 2022-02-08; First posted 2022-03-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-09

CONDITIONS: Medial Patellofemoral Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Poly-Tape Devices: Poly-Tape Devices for Medial Patellofemoral Ligament (MPFL) Reconstruction
  Interventions: Device: Poly-Tape Devices

INTERVENTIONS:
Device: Poly-Tape Devices — Poly-Tape Devices, 10mm Poly-Tape or 5mm Infinity-Lock Tape, for Medial Patellofemoral Ligament (MPFL) Reconstruction
  Other Names: 10mm Poly-Tape; 5mm Infinity-Lock Tape

SUMMARY:
This is a Post Market Clinical Follow Up Study in Orthopaedics. It will verify the long-term safety and performance of the device in the intended patient population, when indicated for the reconstruction of a ligament in the kneecap - the Medial Patellofemoral Ligament (MPFL).

The Medical Devices in this study, 10mm Poly-Tape and 5mm Infinity-Lock Tape, are Class III CE-Marked devices manufactured by Xiros Ltd. Both devices fall under the Poly-Tape family. Poly-Tapes are single-use devices, they are indicated for patients requiring soft tissue approximation and reconstruction of ligaments and tendons. The device can be fixed to the bone using several different methods, including screws.

This study is a prospective, multicentre, consecutively recruited non-randomised study. The total length of the study is expected to be 7 years. This includes a recruitment period of approximately 24 months and a 5-year follow-up. A total of 55 subjects will be enrolled into the study with follow up at 6 months, 1 year, 2 years and 5 years in clinic and by questionnaires. All subjects treated with either the 10mm Poly-Tape or 5mm Infinity-Lock Tape for MPFL reconstruction, will be consecutively recruited into the study.

ELIGIBILITY:
Inclusion Criteria:

Patient must be 13 years old or above. Patients who require MPFL reconstruction. Patients willing to participate in the study and have been informed of the nature of the study, agree to its follow-up and have provided written informed consent as approved by the Research Ethics Committee (REC).

Exclusion Criteria:

These devices should not be used in procedures which bridge, disturb, or disrupt the growth plate in immature patients since they will not elongate as the patient grows.

Patients known to be hypersensitive to titanium alloy or polyester. Appropriate tests should be carried out on patients with suspected material sensitivity prior to implantation.

Patients with any infections or structural or pathological condition of the bone or soft tissue that would be expected to impair healing or secure fixation. Bone quality should be assessed prior to surgery.

Patients who are unable or unwilling to restrict activities to prescribed levels or to follow the rehabilitation instructions during the healing period.

Patients for whom the implantation is intended to be non-permanent, since they integrate well with the patient's tissue.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who require MPFL reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Kujala Score | 1 year
  The primary performance objective is to determine the effect of MPFL reconstruction on symptoms and functional limitations 1 year after surgery, measured using the Kujala .Total score. Total scores range from 0 to 100 with high scores indicating good
Redislocation/subluxation events | 1 year
  The primary safety objective is to assess redislocation/subluxation events at 1 year after surgery

SECONDARY OUTCOMES:
Full range of motion (ROM) | 5 years
  Secondary performance objectives are to determine the effect of MPFL reconstruction on the following during the performance lifetime of the device: Full range of motion (ROM)
Norwich Patellar Instability (NPI) score | 5 years
  Change from baseline Norwich Patellar Instability (NPI) score at each visit up to 1 year. The score is made up of 0 to 250. Out of the total score-able answers, where "don't do" answered questions are deducted, the total score is then converted as a percentage based on the number of scored responses provided. A higher percentage indicate higher severity of patellar instability
Patient-reported quality of life (RANDShort form 36) | 5 years
  Secondary performance objectives are to determine the effect of MPFL reconstruction on the following during the performance lifetime of the device: Patient-reported quality of life 0-100 a higher sore indicates a higher health state
Patient-reported activity levels | 5 years
  Secondary performance objectives are to determine the effect of MPFL reconstruction on the following during the performance lifetime of the device: Patient-reported activity levels 0-10 , 10 is a high level of activity
Patient satisfaction with Surgery | 5 years
  Secondary performance objectives are to determine the effect of MPFL reconstruction on the following during the performance lifetime of the device: Patient satisfaction with Surgery.
  Yes or No
Adverse events, including re-dislocation/subluxation | 5 years
  Secondary safety objectives include: Adverse events, including

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - Tameside and Glossop Integrated Care NHS Foundation Trust, Manchester
  - University of North Midlands NHS Trust, Stoke-on-Trent
  - Hampshire Hospitals NHS Foundation Trust, Winchester
  - Somerset NHS Foundation Trust, Yeovil

IPD SHARING:
Plan to Share IPD: No